CLINICAL TRIAL: NCT05178576
Title: A Single Arm Phase II Study to Evaluate Treatment With Gevokizumab in Patients With Stage II/III Colon Cancer Who Are ctDNA-positive After Curative Surgery and Adjuvant Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug not available for the study duration.
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Novartis Pharmaceuticals (Industry); Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FC-12
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Colon Cancer
Keywords: ctDNA positive; adjuvant; Signatera; gevokizumab; chemotherapy; Stage II; Stage III; Microsatellite Stable (MSS)
MeSH Terms: conditions — Colonic Neoplasms | interventions — gevokizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Arm 1 (Experimental): ctDNA positive Gevokizumab for 1 year (maximum of 13 cycles)
  Interventions: Drug: Gevokizumab; Diagnostic Test: Signatera test

INTERVENTIONS:
Drug: Gevokizumab — 120mg IV on day 1 of every 28-day cycle for 1 year (maximum of 13 cycles)
Diagnostic Test: Signatera test — ctDNA monitoring at weeks 8, 12, 24, 36, 48, 60 and 72 unless disease recurrence is documented.

SUMMARY:
This study will look at the recurrence-free survival of microsatellite-stable (MSS) colon cancer in patients are ctDNA (circulating tumor DNA) positive and treated with gevokizumab.

DETAILED DESCRIPTION:
NSABP FC-12 is a single-arm, multi-centered phase II study to evaluate recurrence-free survival in patients with stage II/III microsatellite-stable (MSS) colon cancer who have undergone curative surgery, adjuvant chemotherapy, are ctDNA (circulating tumor DNA)-positive and treated with gevokizumab.

Patients with stage III resected MSS colon cancer (CRC) who are less than or equal to (≤) 6 weeks after completion of at least 3 months of a standard adjuvant chemotherapy regimen, who are interested in participating in the FC-12 study are eligible for pre-entry ctDNA testing for ctDNA-positivity using the Signatera™ assay via the FC-12 study. Within 6 weeks after completion of adjuvant therapy, stage III patients who have signed the FC-12 Pre-Screening ctDNA consent will have blood and primary tissue samples collected and submitted to Natera for ctDNA evaluation. Commercial ctDNA assay results will not be accepted for study entry. For 150 patients screened in this CRC population, the ctDNA-positivity rate is expected to be approximately 20%.

Note: Patients with stage II MSS colon cancer who were determined to be ctDNA-positive by Natera's Signatera™ commercial assay (i.e., outside of the study) after curative resection may be considered for ctDNA confirmation of ctDNA-positivity via the FC-12 study provided that all the following are met:

* The patient has completed of at least 3 months of a standard adjuvant chemotherapy regimen.
* ctDNA samples will be collected and submitted for ctDNA-positivity confirmation by the Signatera™ assay via the FC-12 study within ≤ 8 weeks after the patient has completed adjuvant chemotherapy.
* The patient otherwise meets eligibility criteria. And,
* the patient will be able to start study therapy within 14 weeks after completion of adjuvant chemotherapy.

All eligible consenting patients who have ctDNA-positivity confirmed via the FC-12 study must begin study therapy within 14 weeks from the completion of adjuvant chemotherapy. Patients will receive gevokizumab (120mg IV) on Day 1 of every 28-day cycle for a maximum of 1 year (e.g., 13 cycles: 1 cycle = 28 days). Patients will continue to receive 13 cycles (1 year) of study therapy unless the patient elects to discontinue study medication, does not adhere to the study per the investigator, experiences intolerable drug toxicity, or has disease recurrence confirmed by imaging.

ctDNA will be monitored at Weeks 8, 12, 24, 36, 48, 60, and 72 unless disease recurrence is documented by imaging. Imaging will include CT scan of chest, abdomen and pelvis and will occur every 24 weeks (6 months) for the duration of the patient's participation in the study or until imaging confirms recurrence.

All patients will be followed for approximately 18 months after initiating study therapy or until imaging confirms recurrence whichever comes first.

The sample size and maximum enrollment for this single arm phase II trial is approximately 31 patients with stage II patient accrual capped at no more than 8 patients. Enrolled patients who withdraw consent prior to receiving study therapy or who are unable to begin study therapy will be replaced.

Safety assessments will occur at intervals per protocol (Section 5.0). Drug toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE 5.0).

Submission of archived tumor tissue and blood for FC-12 correlative science studies will be a requirement for all patients enrolled into the study. Serial blood samples will be collected at specified time points throughout the study for gevokizumab pharmacokinetics (PKs) and anti-drug antibody (ADA) assessment.

Stool samples for FC-12 correlative science microbiome studies are optional.

ELIGIBILITY:
Inclusion Criteria:

The ECOG performance status must be 0 or 1.

Patients must have histologically/pathologically confirmed stage II/III adenocarcinoma of the colon (per AJCC 8th edition) with R0 resection by open laparotomy or laparoscopic-assisted colectomy.

There must be documentation by CT scan with contrast that the patient has no evidence of measurable metastatic disease including assessment of chest, abdomen, and pelvis. (Note: MRI will be accepted for patients unable to have CT scans with contrast.)

Patients must have completed at least 3 months of a standard adjuvant chemotherapy regimen.

The distal extent of the tumor must be greater than or equal to 12 cm from the anal verge on colonoscopy or above the peritoneal reflection as documented during surgery or on pathology specimen.

Patients with microsatellite stable (MSS) proficient mismatch repair (pMMR) tumors are eligible.

Patients must be ctDNA-positive as determined by the Natera Signatera™ assay from samples submitted to Natera within less than or equal to 6 weeks after completing adjuvant chemotherapy. The study will provide pre-entry ctDNA testing for consenting stage III patients. Note: Stage II colon cancer patients may be ctDNA tested via the FC-12 study provided all the following criteria are met:

* The patient must have been previously determined to be ctDNA-positive by Natera's Signatera™ commercial assay outside of the study (i.e., at the time of resection).
* The patient has received at least 3 months of a standard chemotherapy regimen.
* Patients must sign the FC-12 ctDNA Screening consent and samples must be submitted to Natera within less than or equal to 6 weeks after completion of the adjuvant chemotherapy for reconfirmation of ctDNA-positivity by the Signatera™ assay via the FC-12 study.

Patients must be able to begin study therapy within 14 weeks after the completion of adjuvant chemotherapy.

At the time of study entry, blood counts performed within 2 weeks prior to study entry must meet the following criteria:

* ANC must be greater than or equal to 1500/mm3,
* Platelet count must be greater than or equal to 100,000/mm3; and
* Hemoglobin must be greater than or equal to 9 g/dL. (Note: transfusions maybe used to correct hemoglobin for patients experiencing anemia from therapy who otherwise would be eligible for the study.)
* Albumin greater than 3.0 g/dL

The following criteria for evidence of adequate hepatic function performed within 2 weeks prior to study entry must be met:

* Total bilirubin must be less than or equal to 1.5 x ULN. (Note: any elevated bilirubin has to be asymptomatic.)
* AST and ALT must be less than or equal to 3.0 x ULN for the lab. (Note: In patients with elevated ALT or AST, the values must be stable for at least 2 weeks and with no evidence of biliary obstruction on imaging.)

Creatinine must be less than or equal to 3.0 x upper limit of normal (ULN).

All chemotherapy toxicities (excluding alopecia and amenorrhea) must be less than grade 2 at the time study therapy is to begin.

Patients must have no evidence of opportunistic infections.

Female patients of childbearing potential must have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Male and female patients with reproductive potential must agree to use accepted effective methods of contraception while receiving study therapy and for at least 90 days (3 months) after the completion of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

Diagnosis of anal or small bowel carcinoma.

Colon cancer other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.

Patients with MSI-high defective mismatch repair (dMMR) tumors are ineligible.

An elevated CEA above institutional normal value. For smokers a higher institution ULN is acceptable.

Use and/or receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, monoclonal anti-bodies) or radiation therapy within 4 weeks prior to receiving first dose of study therapy.

Persistent diarrhea greater than grade 1.

History of active or latent tuberculosis (TB) infection. If presence of TB (active or latent) is established, then treatment for TB must be completed according to local guidelines prior to the screening.

Active untreated or uncontrolled systemic fungal, bacterial or viral infections, or active infection requiring systemic anti-infectious therapy.

Current or history of systemic autoimmune disease requiring systemic immunosuppressive therapy will not be allowed. Note: the following will not be exclusionary: 1) the presence of laboratory evidence of autoimmune disease (e.g. positive antinuclear antibody titer or lupus anticoagulant) without associated symptoms; 2) clinical evidence of vitiligo or other forms of depigmenting illness; 3) mild autoimmunity not impacting the function of major organs (e.g. controlled Hashimoto thyroiditis, limited psoriasis).

Patients will be excluded if they are on systemic steroid therapy that cannot be discontinued (except for the use of prednisone or equivalent less than 0.125mg/kg/day as replacement therapy). Inhaled or topical steroids are permitted.

Receipt of live attenuated vaccination within 30 days prior to study entry.

Active or chronic hepatitis B virus (HBV) or hepatitis C virus (HCB) infections.

Note: Patients with a history of hepatitis C virus (HCV) infection must have been treated and with confirmation of cure, can be eligible.

Active infection or chronic infection requiring chronic suppressive antibiotics.

History of allogeneic organ or bone marrow transplantation.

Any of the following cardiac conditions:

* documented NYHA Class III or IV congestive heart failure,
* symptomatic arrhythmia.
* History of myocardial infarction (MI), angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to starting study treatment
* Clinically significant cardiac arrhythmias
* Uncontrolled congestive heart failure Active documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).

Major surgical procedure within 28 days prior to study entry.

Other malignancies: unless the patient is considered disease-free and has completed therapy for the malignancy greater than or equal to 12 months prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, and basal cell and squamous cell carcinoma of the skin. Other in situ neoplasms will be reviewed by the Protocol Officer and/or Protocol Chair.

Psychiatric or addictive disorders or other conditions that in the opinion of the investigator would preclude the patient from meeting the study requirements or interfere with interpretation of study results.

Pregnancy or lactation at the time of study entry.

Use of any investigational agent within 4 weeks prior to the first dose of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) at one year | From the initiation of study therapy through 1 year of follow-up
  Percentage of patients alive absent recurrence

SECONDARY OUTCOMES:
Clearance of ctDNA | From the initiation of study therapy to 8 weeks
  Percentage of patients who have converted to negative ctDNA assay at 8 weeks from start of study therapy
Duration of Recurrence-free survival (RFS) with ctDNA clearance at 8 weeks from start of study therapy | From the initiation of study therapy through 1 year of follow-up
  Percentage of patients who have converted to a negative ctDNA assay at 8 weeks and are absent recurrence at one year
Duration of Recurrence-free survival (RFS) without ctDNA clearance at 8 weeks | From the initiation of study therapy through 1 year of follow-up
  Percentage of patients who have not converted to a negative ctDNA assay at 8 weeks and are absent a recurrence at one year.
Frequency of adverse events assessed using CTCAE 5.0 | From beginning of study therapy until 90 days after last dose, approximately 15 months
  Distribution of patients (percentage) by maximum observed grade of adverse event (0-5).
Serum concentration | From beginning of study therapy until 30 days after last dose
  Describe serum concentration (pharmacokinetics) of gevokizumab
Immunogenicity | From beginning of study therapy until 30 days after last dose
  Describe anti-drug antibodies to gevokizumab

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (5):
- United States (5):
  - UF Health Davis Cancer Pavilion and Shands Med Plaza, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - AHN Cancer Institute, Pittsburgh, Pennsylvania